CLINICAL TRIAL: NCT07103902
Title: Effects of Aerobic Exercise on Obsessive-Compulsive Disorder Symptoms and Cognitive Flexibility
Brief Title: Aerobic Exercise and Obsessive-Compulsive Disorder Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Thomas Adams, PhD, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000040629
Record Dates: First submitted 2025-07-24; First posted 2025-08-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-07

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: Anxiety Disorders; Mental Disorders; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Exercise (Experimental)
  Interventions: Behavioral: Moderate-Intensity Exercise
- Low-Intensity Exercise (Other): Control
  Interventions: Behavioral: Low-Intensity Exercise

INTERVENTIONS:
Behavioral: Moderate-Intensity Exercise — Participants will engage in 20 minutes of cycling at approximately 70% max heart rate with a 2.5 minute warm up and a 2.5 minute cool down.
  Arms: Moderate-Intensity Exercise
Behavioral: Low-Intensity Exercise — Participants will engage in 20 minutes of cycling at approximately 40-50% max heart rate with a 2.5 minute warm up and a 2.5 minute cool down.
  Arms: Low-Intensity Exercise

SUMMARY:
The purpose of this study is to examine the acute effects of exercise on cognitive flexibility and symptom reactivity. The main questions it aims to answer are:

Does moderate intensity physical activity reduce subjective distress, compulsive urges, and intrusions- and increase cognitive flexibility- in adults with obsessive-compulsive disorder compared to low-intensity physical activity?

Researchers will compare low- to moderate-intensity exercise to see if moderate physical activity increases cognitive flexibility and reduces symptom reactivity in adults with obsessive-compulsive disorder (OCD).

Participants will:

Complete self-report surveys, psychiatric interviews, and cognitive tasks.

Be assigned to either a low- or moderate-intensity exercise condition and complete physical activity.

Repeat cognitive and symptom measures following the exercise intervention.

DETAILED DESCRIPTION:
The proposed study aims to determine if moderate physical activity increases cognitive flexibility (aim 1) and reduces symptom reactivity (aim 2) in adults with obsessive-compulsive disorder (OCD).

Adults with obsessive-compulsive disorder (OCD) will be asked to participate in this study, which consists of two visits in addition to a self-report survey between these two visits.

This study will randomize 50 adults with obsessive-compulsive disorder (OCD) for aims 1 and 2.

First, participants will complete a phone screen to determine preliminary eligibility. During Session 1, participants will be consented and complete the diagnostic interview for anxiety, mood, and obsessive-compulsive related disorders (DIAMOND), the baseline probabilistic reversal learning (PRL) task, the symptom reactivity task, and self-report measures in-person. Between sessions 1 and 2, participants will be asked to complete several self-report measures via RedCap survey link.

Session 2 will take place 7-10 days following Session 1. Upon arrival to the lab, participants will be randomized (1:1) to a moderate-intensity physical activity or a low-intensity control condition. Randomization will be stratified based on sex and age to minimize demographic differences. Participants will be blind to allocation.

Individuals assigned to the moderate-intensity physical activity condition will engage in 20 minutes of cycling at approximately 70% max heart rate with a 2.5 minute warm up and a 2.5 minute cool down. In the low-intensity control condition, participants will cycle for 20 minutes at a 40-50% max heart rate with a 2.5 minute warm up and a 2.5 minute cool down. Participants will be instructed to maintain pedaling speed within ranges appropriate for each condition (e.g., 30-40 RPM for low-intensity) and research staff will adjust resistance level throughout the session to ensure that they stay within the target heart rate zones. Participants will be asked to rate their perceived exertion at five minute intervals throughout the session.

Following moderate- or low-intensity exercise, participants will complete follow-up administrations of cognitive flexibility and symptom reactivity tasks.

Cognitive flexibility will be assessed using the computerized Lucky Picture Selection Game, a probabilistic reversal learning (PRL) task. Participants choose between three images to earn points for a monetary bonus, with one image being the "lucky picture." The task includes ~260 trials across low and high volatility blocks, reflecting reversal frequency.

Symptom reactivity will be assessed using the The Braga Obsessive Compulsive Symptom Image Set (BOCI), an open-source, validated task designed to provoke obsessive-compulsive disorder (OCD) symptoms across washing, checking, and symmetry symptom dimensions.

Exercise intensity will be measured as a function of maximum heart rate. A PolarTech chest-strap heart rate monitor will be used during the exercise/control conditions to maintain the target intensity level. Heart rate will be monitored continuously throughout the session.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 to 64 years
* Meet diagnostic criteria for OCD (per the DIAMOND)
* Stable psychiatric or medication treatment (if ≥4-weeks), or if no active treatment. Psychotropic medications will be reviewed with the study psychiatrist on a case by case basis.

Exclusion Criteria:

* Active or unmanaged psychotic disorders, pervasive developmental disorders, bipolar disorder, current substance use disorder (moderate-to-severe), or high risk for suicide (defined as attempt, plan, or intent within past 3 months)
* Documented motor impairments and medical condition(s) that prohibit physical exercise
* Those who are pregnant or trying to become pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive flexibility will be assessed using a probabilistic reversal learning (PRL) task called the Lucky Picture Selection Game. | Cognitive flexibility will be initially measured on day 1. Follow-up administrations will be completed 7-10 days later after the exercise intervention during session 2.
Symptom reactivity will be assessed using the Braga Obsessive Compulsive Symptom Image Set (BOCI). | Symptom reactivity will be initially measured on day 1. Follow-up administrations will be completed 7-10 days later after the exercise intervention during session 2.
Exercise intensity will be measured using a PolarTech chest-strap HR monitor. | Exercise intensity will be measured during 7-10 days after baseline, during session 2.
  Exercise intensity will be measured as a function of maximum heart rate (70% Max HR for moderate intensity condition and 40-50% max heart rate for low intensity condition).

CONTACTS AND LOCATIONS:
Locations (1):
- Temple Medical Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw, de-indentified data.
Time Frame: IPD will be shared within one year of study completion.
Access Criteria: Access to IPD will be made available upon request.